CLINICAL TRIAL: NCT05892406
Title: 3 Dimensional Accuracy of Dental Implant Placement: Randomised Controlled Trial Comparing Robotic Assistance, Dynamic Navigation, and Static Guide
Brief Title: Accuracy of Dental Implant Position Robotic Assistance, Dynamic Navigation, or Static Guide?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Maurizio Tonetti, Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH9H-2023-T109
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Dental Implant
Keywords: robotic surgery; dynamic surgical navigation; 3D printed static guide; Accuracy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Static guide (Active Comparator): Prosthetically guided Implant placement utilising a 3D printed static guide based on a digital plan
  Interventions: Device: Static guide
- Dynamic navigation (Active Comparator): Prosthetically guided Implant placement utilising a dynamic navigation system based on a digital plan
  Interventions: Device: Dynamic navigation
- Robotic system (Experimental): Prosthetically guided Implant placement utilising robotic surgery based on a digital plan
  Interventions: Device: Robotic system

INTERVENTIONS:
Device: Static guide — A static guide will be designed and fabricated based on CBCT and intra-oral scan. Implant will be placed under the assistance of statistic guide through the whole procedure.
  Arms: Static guide
Device: Dynamic navigation — Implant will be placed under the assistance of dynamic navigation.
  Arms: Dynamic navigation
Device: Robotic system — Implant will be placed under robotic arm and human collaboration.
  Arms: Robotic system

SUMMARY:
For free hand dental implant placement, a key difficulty is to accurately control the position. Improving precision of dental implant placement is considered important for safety and efficacy of tooth replacement with dental implants. There are 3 available methods to improve implant position according to a digitally constructed prosthetically guided plan: the use of a 3D printed static guide, the use of a dynamic navigation system or the use of a robotic system. The goal of this randomized controlled trial is to compare the positional implant accuracy, the surgical time, and patient satisfaction among three methods of digital guidance: the use of a 3D printed static guide, dynamic navigation, and robotic assisted surgery. Patients requiring single tooth replacement with a dental implant will be digitally planned using a CBCT and an intraoral digital scan. Subjects will be randomized to one of the three treatment modalities based on the plan. The accuracy of placement will be assessed evaluating the difference between the planned and the actual position using a follow-up scan taken at the end of the surgery. Subjects will be followed up for one year to assess both patient reported and professional outcomes.

DETAILED DESCRIPTION:
For free hand dental implant placement, a key difficulty is to accurately control the position. Improving precision of dental implant placement is considered important for safety and efficacy of tooth replacement with dental implants. There are 3 available methods to improve implant position according to a digitally constructed prosthetically guided plan: the use of a 3D printed static guide, the use of a dynamic navigation system or the use of a robotic system. The goal of this randomized controlled trial is to compare the positional implant accuracy, the surgical time, and patient satisfaction among three methods of digital guidance: the use of a 3D printed static guide, dynamic navigation, and robotic assisted surgery. Patients requiring single tooth replacement with a dental implant will be digitally planned using a CBCT and an intraoral digital scan. Subjects will be randomized to one of the three treatment modalities based on the plan. The accuracy of placement will be assessed evaluating the difference between the planned and the actual position using a follow-up scan taken at the end of the surgery. Platform deviation will be measured digitally. Subjects will be followed up for one year to assess both patient reported and professional outcomes and associate them with the precision of implant position.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a single missing tooth, with sufficient bone volume and keratinized tissue at edentulous site, willing to comply with research appointments/schedule.

Exclusion Criteria:

* Pregnancy or intention to become pregnant at any point during the study duration; with any systematic diseases/conditions that are contradictions to dental implant treatment; inability or unwillingness of individual to give written informed consent; inability of follow-up according to the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Implant positional accuracy | Immediately after surgery
  Implant accuracy will be measured as discrepancy between the digital plan and t actual position of the implant.
Peri-implant soft tissue health | 12 month follow-up
  Defined according to the peri-implant health case definition by Berglundh et al 2017 and the ID-COSM international consensus conference

SECONDARY OUTCOMES:
Surgery time | intraoperative
  Time needed for surgery procedure will be recorded from anaesthesia to connection of cover screw/healing abutment.
Pain perception | Immediately after surgery
  Patient pain perception during surgery will be recorded using visual analogue scale (VAS with range from 0 to 10 with 10 being the highest possible pain experience) .
Pain perception | 7 days after surgery
  Patient pain perception after surgery will be recorded using visual analogue scale (VAS with range from 0 to 10 with 10 being the highest possible pain experience) .
Patient preference | Immediately after surgery
  Assessed using a visual analogue scale (VAS, 100 mm, with 0=least desirable option and 100 = most desirable option.
Surgeon preference | Immediately after surgery
  Assessed using a visual analogue scale (VAS, 100 mm, with 0=least desirable option and 100 = most desirable option.
Esthetics of the restoration | 12-months follow-up after delivery of crown
  Assessed using the PES-WES scale as reported by Belser et al. with 0 being the worst and 14 the best value in the scale
Cytokine concentrations in PISF | 12-months follow-up after delivery of crown
  Cytokine concentration in peri-implant sulcus fluid assesed by MULTIPLEX ELISA of IL-1, TNFa, IL-6 with lower concentrations representing less inflammation.
Submarginal microbiome | 12-months follow-up after delivery of crown
  16S assessment of microbiome diversity (Shannon index) with greater diversity representing a more stable microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, PhD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (2):
- China (2):
  - Department of Oral and Maxillofacial Implantology, Shanghai, Shanghai Municipality
  - Shanghai Perio-Implant Innovation Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No